CLINICAL TRIAL: NCT00052689
Title: A Randomized Phase II Trial of PS-341 and Gemcitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Bortezomib With or Without Gemcitabine in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01799; NCI-2012-01799 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N014C; CDR0000258670; N014C (Other: North Central Cancer Treatment Group); N014C (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Duct Cell Adenocarcinoma of the Pancreas; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bortezomib; Gemcitabine

ARMS (2):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Patients with progressive disease crossover to arm II.
  Interventions: Drug: bortezomib
- Arm II (Experimental): Patients receive bortezomib as in arm I and gemcitabine IV over 30 minutes on days 1 and 8.
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bortezomib — Given IV
Drug: gemcitabine hydrochloride — Given IV
  Arms: Arm II

SUMMARY:
Randomized phase II trial to compare the effectiveness of bortezomib with or without gemcitabine in treating patients who have metastatic pancreatic cancer. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bortezomib with gemcitabine may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the objective response rate in previously untreated patients with metastatic pancreatic adenocarcinoma treated with bortezomib with or without gemcitabine.

II. Compare the toxicity of these regimens in these patients. III. Compare the progression-free, 6-month, and overall survival of patients treated with these regimens.

IV. Compare the change in overall quality of life (QOL) and in subcomponents of QOL of patients after treatment with 2 consecutive courses of these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1of 2 treatment arms.

ARM I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Patients with progressive disease crossover to arm II.

ARM II: Patients receive bortezomib as in arm I and gemcitabine IV over 30 minutes on days 1 and 8.

Courses in both arms repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life (QOL) is assessed at baseline and before courses 2 and 4. Patients who crossover to arm II from arm I complete QOL questionnaires before the first 2 courses of arm II therapy.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic ductal or undifferentiated adenocarcinoma consistent with a pancreatic primary for which no standard curative measures exist

  * No locally advanced disease only
* No islet cell, acinar cell, or cystadenocarcinomas
* Measurable disease

  * At least one lesion whose longest diameter can be accurately measured as 2 cm or greater by conventional techniques OR 1 cm or greater by spiral CT scan
  * A tumor lesion in a previously irradiated area allowed provided it is histologically confirmed disease with radiographic progression from a post-radiotherapy CT scan
* No CNS metastasis
* Performance status - ECOG 0-2
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (stents allowed)
* AST no greater than 5 times ULN
* PT and PTT no greater than ULN*
* Creatinine no greater than 1.5 times ULN
* No other prior malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No neuropathy greater than grade 1
* No underlying disease state associated with active bleeding
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* More than 4 weeks since prior biologic therapy or immunotherapy
* No concurrent immunotherapy
* No concurrent colony-stimulating factors during the first course of the study
* No prior gemcitabine (even as a radiosensitizing agent)
* No prior chemotherapy

  * Radiosensitizing agent as adjuvant therapy or for locally advanced disease allowed
* No other concurrent chemotherapy
* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to 25% or more of the bone marrow
* No concurrent radiotherapy
* No prior bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2002-12; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response (CR, PR) rate in 2 consecutive courses within 6 months (Arm I) | Up to 6 months
  An evaluable patient will be classified as a treatment 'success' if they have a confirmed tumor response (CR, PR). The proportion of successes will be estimated by the total number of evaluable patients. 95% confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.
Proportion of patients alive at 6 months (Arm II) | At 6 months
  An evaluable patient will be classified a treatment 'success' if they are alive at 6 months. The proportion of successes will be estimated by the total number of evaluable patients. 95% confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Survival time | Time from randomization to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from randomization to documentation of disease progression, assessed up to 5 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time to treatment failure | Time from the date of randomization to the date at which the patient is removed from the treatment due to progression, toxicity, or refusal, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Alberts, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States